CLINICAL TRIAL: NCT01217190
Title: Open-Label Randomized, Single Oral Dose, Two-Way Crossover Bioequivalence Study Comparing Ondansetron Orally Dissolving Film Strip 8 mg With Zofran Orally Disintegrating Tablets (ODT) (Containing Ondansetron 8 mg) in Healthy Adults
Brief Title: Crossover Study Comparing Ondansetron Orally Dissolving Film Strip (ODFS) With Zofran Orally Disintegrating Tablets
Acronym: 01905/08-09
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MonoSol Rx (Industry)
Responsible Party: Sponsor
Organization: Aquestive Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OND/CR/020/08-09; NCT01216969 (obsolete NCT alias)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Nausea and Vomiting, Postoperative; Nausea With Vomiting Chemotherapy-Induced
Keywords: Bioequivalence, safety, and tolerability
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: Two period study, two treatment, randomized sequence
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron ODFS then Zofran ODT (Experimental): Single dose of Ondansetron Orally Dissolving Film Strip 8 mg followed by single dose of Zofran ODT® Orally Disintegrating Tablet containing Ondansetron 8 mg with 7 days washout between the 2 periods
  Interventions: Drug: Ondansetron (ODFS); Drug: Zofran (ODT)
- Zofran ODT then Ondansetron ODFS (Experimental): Single dose of Zofran ODT® Orally Disintegrating Tablet containing Ondansetron 8 mg followed by single dose of Ondansetron Orally Dissolving Film Strip 8 mg with 7 days washout between the 2 periods
  Interventions: Drug: Ondansetron (ODFS); Drug: Zofran (ODT)

INTERVENTIONS:
Drug: Ondansetron (ODFS) — Test Article
  Other Names: Ondansetron Orally Dissolving Film Strip
Drug: Zofran (ODT) — Comparator
  Other Names: Zofran Orally Disintegrating Tablet

SUMMARY:
This was an open-label, balanced, two-treatment, two-period, randomized sequence crossover bioequivalence study with a 7-day washout between periods. Each treatment was administered after an overnight (10 hours) fast.

DETAILED DESCRIPTION:
This was an open label, balanced, randomized, two-treatment, two-period, randomized sequence crossover study conducted in healthy adult male and female volunteers. Subjects checked into the study center on Day -1 of each study period at least 12 hours prior to dosing on Day 1. Subjects were served dinner between 8:00 pm to 8:30 pm to ensure minimum 10 hours fast prior to dosing in both periods. Subjects received the 2 treatments in a randomized order with a 7-day washout between the 2 periods.

Treatment A: single dose of ondansetron ODFS 8 mg was orally administered, allowed to dissolve, swallowed with saliva, followed with 240 mL room temperature drinking water

Treatment B: single dose of Zofran ODT (containing ondansetron 8 mg) was orally administered, allowed to dissolve, swallowed with saliva, followed with 240 mL room temperature drinking water

ELIGIBILITY:
Inclusion Criteria:

* Volunteer should have written informed consent.
* Volunteer healthy adult within 18-45 years of age (inclusive).
* Body mass index of 18.5 kg/m^2 and 25 kg/m^2, body weight not less than 50 kg.
* Volunteer must be of normal health.
* Volunteer should have a normal ECG, chest X-ray and vital signs.
* If study volunteer is a female and is of child bearing potential practicing an acceptable method of birth control for the duration of the study.

Criteria: Exclusion Criteria:

* Volunteer doesn't understand the informed consent.
* Volunteer with a history of hypersensitivity or idiosyncratic reaction to study drug or any other related drug.
* Volunteer having any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function, by standard laboratory, imaging or monitoring procedures
* Volunteer who smokes regularly, alcohol or drug abuse
* Volunteer who has taken over the counter or prescribed medications
* Volunteer with clinically significant abnormal values of laboratory parameters.
* Volunteer who has participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Female volunteer demonstrating a positive pregnancy screen with urine pregnancy test (strip method).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09-16 (Actual); Primary Completion 2008-09-26 (Actual); Study Completion 2008-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudershan Vishwanath, MD, Principal Investigator — Vimta Labs Ltd.
Locations (1):
- VIMTA VHS Research Centre, Adyār, Chennai, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned sample size was 48. Of the 48 participants enroll in the study, 46 completed the study.
Pre-assignment Details: A total of 68 volunteers (52 males and 16 females) were screened for enrollment and a total of 48 volunteers (41 males and 7 females) were subsequently admitted to the study.
Groups:
- Experimental: Ondansetron ODFS, Then Zofran ODT: Participants first received a single oral dose of Ondansetron Orally Dissolving Film Strip (ODFS) 8 mg after an overnight fast of at least 10 hours. After a washout period of 7 days, they then received a single oral dose of Zofran Orally Disintegrating Tablet (ODT) containing ondansetron 8 mg after an overnight fast of at least 10 hours.
- Experimental: Zofran ODT, Then Ondansetron ODFS: Participants first received a single oral dose of Zofran Orally Disintegrating Tablet (ODT) containing ondansetron 8 mg after an overnight fast of at least 10 hours. After a washout period of 7 days, they then received a single oral dose of Ondansetron Oral Dissolving Film Strip (ODFS) 8 mg after an overnight fast of at least 10 hours.
Period: First Dosing
Arm/Group | Experimental: Ondansetron ODFS, Then Zofran ODT | Experimental: Zofran ODT, Then Ondansetron ODFS
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Second Dosing
Arm/Group | Experimental: Ondansetron ODFS, Then Zofran ODT | Experimental: Zofran ODT, Then Ondansetron ODFS
Started | 24 | 24
Completed | 24 | 22 (Two subjects withdrew for personal reasons (other than adverse event).)
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: A total of 48 subjects were entered into the study. Two did not complete.
Groups:
- Experimental: Ondansetron ODFS, Then Zofran ODT: 24 participants completed treatment with Ondansetron ODSF 8 mg. After a washout period of 7 days, 24 of the 24 participants who completed the first treatment also completed treatment with Zofran ODT 8mg.
- Experimental: Zofran ODT, Then Ondansetron ODFS: 24 participants completed treatment with Zofran ODT 8 mg. After a washout period of 7 days, 22 of the 24 participants who completed the first treatment also completed treatment with Ondansetron ODSF 8 mg
- Total: Total of all reporting groups
Arm/Group | Experimental: Ondansetron ODFS, Then Zofran ODT | Experimental: Zofran ODT, Then Ondansetron ODFS | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All 24 who entered Ondansetron ODSF first, then Zofran ODT arm completed both periods.
  All 24 subjects who entered Zofran ODT first, then Ondansetron ODSF arm completed the first period, 22 of these 24 subjects completed the second period.
  years
    Age | 29.7 (6.08) | 28.7 (5.6) | 29.2 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No subjects dropped out of Organestron ODFS, then Zofran ODT arm. Two subjects dropped out of Zofran ODT, then Oganestron ODFS arm
  Participants
    Female | 4 | 3 | 7
    Male | 20 | 21 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  India | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum Plasma Concentration occurring at Tmax (Time to reach maximum concentration)
Time Frame: 0,0.33,0.67,1,1.33,1.67,2,2.33,2.67,3,4,6,8,10,12,15,18,24 hours
Population: Pharmacokinetic analysis population comprised all subjects who received study drug in both study periods and completed the study. Two of the 24 subjects in the Zofran ODT then Ondansetron ODSF arm did not return for Period 2 for personal reasons other than adverse events (voluntary withdrawal).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ondansetron ODFS: Single dose of Ondansetron Orally Dissolving Film Strip (ODFS) 8 mg
  ODFS:Two-way cross-over study to compare ODFS 8 mg with Zofran Orally Disintegrating Table (ODT) containing ondansetron 8 mg
- Zofran ODT: Single dose of Zofran (Ondansetron) Orally Disintegrating Tablet (ODT) containing ondansetron 8 mg
  Zofran (ODT): Two-way cross-over study to compare ODFS 8 mg with Zofran ODT 8 mg
Arm/Group | Ondansetron ODFS | Zofran ODT
Number analyzed (Participants) | 46 | 46
ng/mL | 37.282 (14.9177) | 41.108 (17.2442)

2. Primary Outcome: AUCt
Description: Area Under Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration
Time Frame: 0,0.33,0.67,1,1.33,1.67,2,2.33,2.67,3,4,6,8,10,12,15,18,24 hours
Population: 46 subjects completed both Treatments. 2 subjects did not return for Period 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Ondansetron ODFS: Single dose of Ondansetron Orally Dissolving Film Strip 8 mg
  Ondansetron (ODS): Two-wy cross-over study to compare ondansetron ODSF with Zofran ODT
- Zofran ODT: Single dose of Zofran ODT® Orally Disintegrating Tablet 8 mg
  Zofran (ODT): Two way cross-over study to compare ondansetron ODSF with Zofran ODT
Arm/Group | Ondansetron ODFS | Zofran ODT
Number analyzed (Participants) | 46 | 46
ng*hr/mL | 216.269 (83.2883) | 239.463 (100.0745)

3. Primary Outcome: AUCinf
Description: Area Under Plasma Concentration-Time Curve From Time Zero to Time Infinity
Time Frame: 0,0.33,0.67,1,1.33,1.67,2,2.33,2.67,3,4,6,8,10,12,15,18,24 hours
Population: 46 subjects completed both periods. 2 subjects did not complete period 2
Measure: Mean (Standard Deviation); unit: nghr/mL
Groups:
- Zofran ODT: Single dose of Zofran (Ondansetron) ODT® Orally Disintegrating Tablets 8 mg
  Zofran (ODT): Two way cross-over study to compare ondansetron ODSF with Zofran ODT
Arm/Group | Ondansetron ODFS | Zofran ODT
Number analyzed (Participants) | 46 | 46
nghr/mL | 225.032 (88.2551) | 250.673 (107.9654)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the full course of the study (approximately 1 month for each treatment arm).
Description: Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- Ondansetron ODFS: Single dose of Ondansetron Orally Dissolving Film Strip (ODFS) 8 mg
  ODFS: Two-way cross-over study to compare ODFS 8 mg with Zofran Orally Disintegrating Tablet (ODT) containing ondansetron 8 mg
- Zofran ODT: Single dose of Zofran Orally Disintegrating Tablet (ODT) containing ondansetron 8 mg
  Zofran ODT: Two-way cross-over study to compare ODFS 8 mg with Zofran ODT 8 mg
Arm/Group | Ondansetron ODFS | Zofran ODT
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 6/24 | 7/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron ODFS (N=24) | Zofran ODT (N=22)
Eosinophil count increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Increased eosinophil count
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1) — Increased AST
Total bilirubin increased (Hepatobiliary disorders) | 0 (0) | 1 (1) — Increased total bilirubin
Alanine aminotransferase increased (Hepatobiliary disorders) | 2 (2) | 2 (2) — Increased ALT
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Decreased platelet count
Lymphocyte count increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Increased lymphocyte count
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cell count increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — WBC count increased
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Upper respiratory tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes